CLINICAL TRIAL: NCT01029210
Title: Temporomandibular Disorders in Climacteric Women: Pain Sensibility, Risk Posed by Systemic Bone Mass and Diagnostic Made by RDC/TMD Compared to MRI (3.0 Tesla)
Brief Title: Temporomandibular Disorders and Osteoporosis
Acronym: TMDOST
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Instituto de Radiologia do Hospital das Clínicas da FMUSP - InRad (Unknown)
Responsible Party: Principal Investigator, Alessandra Pucci Mantelli Galhardo, Dr, University of Sao Paulo
Other Study IDs: CAPPesq 0175/08
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-11

CONDITIONS: Women; Osteoporosis; Osteopenia; Temporomandibular Disorder
Keywords: osteoporosis; temporomandibular disorders; resonance magnetic
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Increased life expectancy has attracted research attention, interested in provide a quality and healthy aging. According to the latest census conducted in 2010 by IBGE, Brazilian population consists of 97,342,162 women, whom estimates 30 million are between 40 and 65 years old, a period that includes the climacteric. Therefore, clinical conditions such as osteoporosis becomes significant, either from public health policy standpoint or in relation to the social aspect, by compromising life quality. Women also suffer more from temporomandibular disorders (TMD) than men, and the beginning of this situation occurs after puberty, with peaks during the reproductive and remission periods after menopause. Female sex hormones involvement in osteoporosis is well established, but their participation in the TMD is still controversial. Thus, this study aims to investigate the role of systemic bone mass in menopausal women as a risk factor for articular TMD, as well as the TMD pain behavior during menopause transition periods (48 to 55 years), postmenopausal (56-65 years) and senescence (65-70 years). Therefore, 100 women attended by the HC - FMUSP Gynecology Division, Climacteric Sector, were clinically evaluated by the Research Diagnostic Criteria for Temporomandibular Disorders (RDC/TMD), used to obtain diagnoses and their associations, as well as to quantify the TMD pain sensitivity degree through the Craniomandibular Index (CMI), both applied by a single examiner. The bone densitometry provided bone mass data of femoral neck and lumbar spine (L1-L4). The RDC/TMD performance as a diagnostic test also was subjected to analysis, considering the 3.0 Tesla magnetic resonance imaging as reference standard, undergoing 30 women, of 100 assessed, in this imaging exam. After analyzing the results, it was shown that the risk posed by osteopenia was 1.33 (IC95% 1.20 - 1.46), with a risk increase of 0.33, while the risk of osteoporosis showed 1.39 (IC95% 1,20 - 1.23 to 1.55), increased by 0.39. Joint diagnoses predominated (68.0%), while 18.0% muscular diagnoses and 14.0% corresponds to the absence of clinically diagnosable conditions, according to the RDC/TMD. The performance of the RDC/TMD to diagnose articular DTM revealed accuracy of 68.0%, sensitivity of 83.0%, specificity 53.0%, pre-test probability of 52.0%, positive predictive value of 60.0 % and negative 74.0%, positive likelihood ratio of 1.77 and negative 0.32. As for the soreness sensibility in TMD, it was found that aging shows a clear tendency towards its reduction (A =- 4.5, p = 0.0324). Then, the study concluded that the decrease in female sex hormones, peculiar to aging, increases the risk of articular TMD, although this pain disfunction decreases with age. The RDC/TMD can be used for large populations screening, but its indication in clinical practice should be done with caution.

DETAILED DESCRIPTION:
Osteoporosis and temporomandibular disorders are diseases which attack mainly women. Then, this research aims at if if they are related.

ELIGIBILITY:
Inclusion Criteria:

* women
* age between 48 and 70 years old
* densitometry bone actual

Exclusion Criteria:

* diabetes
* fibromyalgia
* lupus, psoriases
* rheumatic disease

Ages: 48 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients attended by the discipline of gynecology - outpatient clinic of climatério
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Galhardo, Principal Investigator — University of Sao Paulo

REFERENCES:
- [Derived] Galhardo AP, da Costa Leite C, Gebrim EM, Gomes RL, Mukai MK, Yamaguchi CA, Bernardo WM, Soares JM Jr, Baracat EC, Gil C. The correlation of research diagnostic criteria for temporomandibular disorders and magnetic resonance imaging: a study of diagnostic accuracy. Oral Surg Oral Med Oral Pathol Oral Radiol. 2013 Feb;115(2):277-84. doi: 10.1016/j.oooo.2012.10.020. PMID 23312922
- See also: Related Info — http://www.teses.usp.br/teses/disponiveis/23/23150/tde-18062011-102133/pt-br.php